CLINICAL TRIAL: NCT06016686
Title: Microelectrode Recordings From the Vagus Nerve in Awake Humans
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VNS
Record Dates: First submitted 2023-07-10; First posted 2023-08-30 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VNS (Experimental): participants with surgically implanted VNS electrodes to treat drug-resistant epilepsy
  Interventions: Other: VNS stimulation and intraneural recordings
- non-VNS participants (Experimental): participants without implanted VNS devices
  Interventions: Other: Record multi-unit activity from intraneural sites

INTERVENTIONS:
Other: VNS stimulation and intraneural recordings — A minimum of three stimulation frequencies (1, 10 and 30 Hz), each up to 60s in duration, will be delivered via the VNS device. Intraneural recordings proximal or distal to the VNS electrodes during delivery of VNS will be performed. Approximately two to five fascicles will be explored in each nerve.
  Arms: VNS
Other: Record multi-unit activity from intraneural sites — Perform a more detailed vagal nerve mapping study by recording from single nerve fibers, including those fibers supplying the heart, lungs, airways and other end-organs. The investigators shall perform functional mapping of the left and right vagus nerves, such as those with cardiac-related and/or respiratory-related neural activity. The research team will also record activity from other nearby fibers to map the differences in neurological behavior in fascicles that control the heart, lungs, airways and other systems.
  Arms: non-VNS participants

SUMMARY:
This Anchillary project uses a refined technique of ultrasound-guided microneurography of the human cervical vagus nerve, an approach developed by Professor Vaughan Macefield and used safely to-date in 44 prior study participants.

The overall goal of this project is to build upon prior data obtained using this approach by undertaking a detailed neurophysiological investigation of the human vagus nerve and to identify the nerve fibers activated during vagal nerve stimulation (VNS) in participants with implanted VNS devices in response to different stimulation parameters. In addition to providing data in unprecedented detail into the physiology of the human vagus nerve, this project will investigate different stimulus intensities, durations and frequencies that differentially excite myelinated and unmyelinated nerve fibers. These results will inform the CSP and guide future development of novel neural interfaces for VNS for various clinical applications.

ELIGIBILITY:
Inclusion Criteria:

* The participant is greater than or equal to (≥)18 years and is less than or equal to (≤) 40 years of age
* English speaking
* Medicare covered or equivalent health insurance from a partner country

Exclusion Criteria:

* Pregnant
* Smokes and is unwilling to abstain from smoking on the day of the experiment.
* Inability or unwillingness to provide written informed consent.
* Individuals with difficulty standing unassisted for 5 minutes during the tilt-table testing
* Individuals found to have a significant carotid artery plaque or intima-media thickness > 1 mm as assessed by ultrasonography during the ultrasound-screening steps of the study visit
* Vagus nerve not visible on ultrasound
* VNS electrodes are not in a suitable location to allow for microelectrode insertion
* Any other clinical reasons deemed by the investigators

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
identify action potential morphology of specific fibers activated by vagal nerve stimulation (VNS) | 4 hours
  assessing vagal nerve activity in epilepsy participants during and in the absence of stimulation. Labchart; spike histogram module
identify ratio of myelinated fibers in specific fibers activated by vagal nerve stimulation (VNS) | 4 hours
  assessing vagal nerve activity in epilepsy participants during and in the absence of stimulation. Labchart; spike histogram module. Whether a nerve fiber is (un)myelinated can be determined by visual inspection. Myelinated fibers typically produce "a positive-going narrow spike profile.
physiological identification of the specific fibers activated by vagal nerve stimulation (VNS) | 4 hours
  assessing vagal nerve activity in epilepsy participants during and in the absence of stimulation. Labchart; spike histogram module. use of tracing and nerve recordings analysis to identify the types of nerves
identify firing rates of the specific fibers activated by vagal nerve stimulation (VNS) | 4 hours
  assessing vagal nerve activity in epilepsy participants during and in the absence of stimulation. Labchart; spike histogram module. in Hertz
identify stimulus current required to activate specific fibers activated by vagal nerve stimulation (VNS) | 4 hours
  assessing vagal nerve activity in epilepsy participants during and in the absence of stimulation. Labchart; spike histogram module. in milli-amps
differences in firing rates of cardiac parasympathetic vagal activity | 4 hours
  compare any changes in parasympathetic vagal activity with participants who have not been implanted with a vagal nerve stimulator (Non-VNS Participants).
  Labchart; spike histogram module. Unit: Hz.
Discharge variability of cardiac parasympathetic nerve fibers | 4 hours
  Vagal nerve stimulator device. Coefficient of variation, %

CONTACTS AND LOCATIONS:
Overall Officials: Vaughan G Macefield, PhD, Principal Investigator — Monash University; John Osborn, Principal Investigator — University of Minnesota
Locations (2):
- University of Minnesota, Minneapolis, Minnesota, United States
- 99 Commercial Road, Prahan Victoria, Australia